

SF\_STAIT001\_ver 2\_Eng Approval Date 18 July 2017

# P16-253 (CITRIN)\_STATISTICAL ANALYSIS PLAN\_FINAL 2.0\_16 Mar 2018

Protocol Number: P16-253 (CITRIN)

Protocol Title: Real world evidence study of the effectiveness of Paritaprevielr -

Ombitasvir + Dasabuvir without Ribavirin in patients with chronic HCV Gt1b infection and compensated liver cirrhosis in the Russian Federation

an observational, multi-center study

SAP version: Final 2.0

Effective date: 19 Mar 2018



## REVISION HISTORY

| No Version | Date | Changes |
|---|---|---|
| 1 1.0 | 16.08.2017 | New Document |
| | | 1) section 9 and corresponding tables shells was updated. |
| | | - additionally to efficiency endpoints the following |
| | | virologic outcomes were added to the analysis:<br>breakthrough, failure to suppress and premature study |
| | | drug discontinuation with no on-treatment virologic |
| | | failure; |
| | | - due to the fact that in the Russian clinical practice tests |
| | | for HCV RNA often have limit of detection higher than |
| | | 50 IU/mL and may vary across laboratories, the |
| 2 2.0 | 16.03.2018 | definitions for effectiveness outcomes were adjusted; |
| | | - additional frequency tables for patients in subgroup |
| | | without missing SVR12 data category were added; |
| | | - method of 95% confidence interval calculation for odds |
| | | ratio in logistic regression analysis was specified; |
| | | 2) the information about time windows for clinical laboratory |
| | | data was moved to section 4.1 "General study design and plan"; |
| | | 3) tables shells for demographics and baseline characteristics |
| | | was changed: one table was divided into several tables; |
| | | 4) list of tables, figures and listings was added |



## TABLE OF CONTENTS

| Abbreviations and definitions | |
|---|---|
| Introduction | Ch |
| Study objectives and variables | Ch |
| 3.1 Study objectives | S |
| 3.2 Variables | 6 |
| Study design | 6 |
| 4.1 General study design and plan | 6 |
| 4.2 Sample size | ~1 |
| 4.3 Randomization and blinding | 00 |
| 4.4 Planned analyses | $\sim$ |
| General considerations | 00 |
| 5.1 Reference start date/time, study day, baseline Error! Bookmark not define | ~ |
| Error! | ~ |
| Analysis populations | 00 |
| Statistical considerations | 9 |
| 7.1 Standard descriptive statistics | 9 |
| 7.2 Statistical tests and common calculations | $\circ$ |
| 7.3 Missing data | |
| 7.4 Multicenter studies | |
| 7.5 Multiple comparisons | $\circ$ |
| Summary of study data1 | |
| 8.1 Subject disposition1 | |
| 8.2 Protocol deviations | |
| 8.3 Demographic and baseline variables1 | _ |
| 8.4 Concurrent illnesses and medical conditions1 | N |
| 8.5 Prior and concurrent medications | N |
| Effectiveness analysis1 | N |
| Safety analysis 1 | S |
| 10.1 Exposure | S |
| 10.2 Adverse events | 6 |
| 10.3 Pregnancies | 6 |
| 10.4 Clinical laboratory evaluations | 6 |
| 10.5 Other safety measures | $\sim$ |
| Pharmacokinetics1 | 00 |
| Other analyses | 00 |
| Interim analyses and data monitoring1 | 00 |
| Technical details and reporting conventions1 | 00 |
| Summary of changes to the Protocol1 | 00 |
| References1 | 9 |
| Tables shells | ÌΔ |
| | viations and definitions viations and variables Study objectives and variables Variables Variables Variables Variables Variables Sample size Randomization and blinding Reference start date/time, study day, baseline Fror! Bookmark not define Windowing conventions It cal considerations It cal considerations Multicenter studies Multicenter studies Multicenter studies Multipe comparisons Subject disposition Protocol deviations Demographic and baseline variables Concurrent illnesses and medical conditions Prior and concurrent medications Prior and concurrent medications Prior and concurrent medications Prior and concurrent medications Prior and concurrent medications Prior and concurrent medical conditions Prior and concurrent medical conditions Prior and concurrent medications Prior and concurrent medical conditions Prior and concurrent medical conditions Prior and concurrent medical conditions Prior and concurrent medical conditions Prior and concurrent medical conditions Pregnancies Adverse events Adverse events Other safety measures Other safety measures Other safety measures It all the protocol It all th |



## 1 Abbreviations and definitions

The abbreviations and the definitions used in this document are listed below.

| Abbreviation | Abbreviation in Full |
|----------------|---------------------------------------------|
| ABBVIE REGIMEN | $Paritaprevir/r - Ombitasvir \pm Dasabuvir$ |
| AE | Adverse event |
| ATC | Anatomical therapeutic chemical code |
| BL | Baseline |
| BMI | Body mass index |
| CHC | Chronic hepatitis C |
| CI | Confidence interval |
| CRF | Case report form |
| CSR | Clinical study report |
| DMC | Data monitoring Committee |
| eCRF | Electronic CRF |
| EoT | End of treatment |
| ICH | International conference on Harmonisation |
| IL28B | Interleukin 28B |
| INR | International normalized ratio |
| IQR | Interquartile range |
| LLoD | Limit of detection |
| LLoQ | Lower limit of quantification |
| PT | Preferred term |
| RBV | Ribavirin |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOC | System organ class |
| SOP | Standard operational procedure |
| SVR | Sustained virological response |
| SVR12 | SVR at 12 weeks after EoT |
| ULoQ | Upper limit of quantification |
| WHO | World Health Organization |
| WHODD | WHO drug dictionary |



### Introduction

Russian Federation (CITRIN). real world evidence study of the effectiveness of Paritaprevir/r - Ombitasvir + Dasabuvir without Ribavirin in patients with chronic HCV Gtlb infection and compensated liver cirrhosis in the This document describes the planned data statistical analysis of an observational, multicenter,

using the Protocol Final version 1.0 dated 29 Nov 2016 and CRF Final version 1.1 dated 16 Mar This SAP is written according to ICH E9 Guideline [1] and Data MATRIX LLC SOP [2]

principal features of the analysis, described in the Protocol, and to include detailed procedures for executing the statistical analysis. The purpose of this document is to provide a more technical and detailed elaboration of the

SAP, explanation will be provided in the clinical study report (CSR). approved SAP may be made prior to database soft lock. In case of deviation from the finalized The SAP needs to be finalized and signed prior to database soft lock. Revisions to the

### S Study objectives and variables<sup>1</sup>

## Study objectives

cirrhosis in a real life setting? ABBVIE REGIMEN without RBV in patients with HCV Gt1b infection and compensated liver The research question of this study is what is the effectiveness of the interferon-free 3DAA

The Protocol defines the following *primary objective* of this study:

to describe the effectiveness of the interferon-free 3DAA ABBVIE REGIMEN without clinical practice. by sustained virological response at 12 weeks after the end of treatment in routine RBV in patients with HCV Gt1b infection and compensated liver cirrhosis as evidenced

The Protocol defines the following secondary objectives of this study:

- to describe the EoT response rate;
- to assess the rate of relapse (timeframe for assessing relapse between EoT and SVR
- cirrhosis treated with AbbVie 3D regimen; to describe baseline characteristics of patients with HCV Gt1b and compensated
- patients in the Russian population; to collect information on co-morbidities and concomitant medications in cirrhotic
- to describe the tolerability of the ABBVIE REGIMEN

<sup>1</sup> This section is based on the sections 8 "Research Question and Objectives", 9.9 "Variables", 9.13.4 "Primary

Effectiveness Endpoints" and 9.13.5 "Secondary Effectiveness Endpoints" of clinical study Protocol.

Page 5 out of 79




### **Variables**

The primary variable of this study (and also effectiveness endpoint) is:

primary effectiveness endpoint. the percentage of patients achieving SVR12 (single last HCV RNA <50 IU/mL 12 weeks [i.e. at least 84 days] after the last actual dose of the ABBVIE REGIMEN) is the

The secondary variables of this study are:

- effectiveness endpoints:
- the percentage of patients with virological response (HCV RNA <50 IU/mL) at EoT;
- the percentage of patients with relapse after EoT (defined as HCV RNA <50~IU/mLat EoT followed by HCV RNA ≥50 IU/mL);
- treatment); one documented HCV RNA <50 IU/mL followed by HCV RNA ≥50 IU/mL during the percentage of patients with relapse during treatment phase (defined as at least
- the number and percentage of patients meeting each and any of the following SVR12 non-response categories:
- relapse during post-treatment phase (defined as HCV RNA <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA >50 IU/mL post-treatment);
- missing SVR12 data and/or none of the above criteria;
- descriptive statistics for baseline characterictics;
- the number and percentage of patients with comorbidities and concomitant medications.
- the number and percentage of patients with adverse events.

### Study design

## General study design and plan<sup>2</sup>

the interferon-free ABBVIE REGIMEN (Paritaprevir/r – Ombitasvir  $\pm$  Dasabuvir) without RBV. This is a post-marketing, prospective, multicenter, observational study in patients receiving

precedes the decision to offer a patient the opportunity to participate in this study. The prescription of a treatment regimen is at the discretion of the physician in accordance with will be offered to participate in this study during a routine clinical visit at the participating sites. with HCV and compensated liver cirrhosis, receiving the interferon-free ABBVIE REGIMEN local clinical practice and label, is made independently from this observational study and This study is focusing on collecting real-world data. Adult patients chronically infected

be taken from medical records. No patient identifiable information will be captured, a unique assessments as recorded in the patient's medical records (source documentation) will be documented in the eCRF. Information for patients enrolled within 2 weeks after initiation of HCV disease characteristics, co-morbidities, co-medication, treatment details, and laboratory written patient authorization form) has been obtained, patient data including demographic data, ABBVIE REGIMEN is collected at routine patient visits therefore baseline patient data should After written Authorization (Consent) for Use/Disclosure of Data form (hereinafter -

<sup>2</sup> This section is based on the sections 9.1 "Study Design" and 9.8 "Description of Activities" of clinical study Protocol.

The EoT time point is included in the analyzed interval.



investigator or designee creates a new patient file. patient number will be automatically allocated by the web based eCRF system once the

routine clinical practice. Follow-up visits, treatment, procedures and diagnostic methods will follow physicians'

between Visit 1 and EoT can be done in case of clinical necessity and physician decision. safety follow-up visit can be done as telephone call contact. Additional observational visits and one 12 weeks follow-up visit (SVR12) after the last dose of ABBVIE REGIMEN. 30 days include at least two observational visits (Visit 1 and EoT) plus one 30 days safety follow-up visit and for up to 12 weeks after treatment completion. 12-week routine treatment regimen will In the study, patients will be observed for the duration of the ABBVIE REGIMEN therapy

study should return to the site to document EoT data. In total, there will be at least four study visits. Patients who prematurely discontinue the

The schedule of the study procedures is presented in table 4.1.

Table 4.1 – Program activities

| Assessment/Procedure | | Treatment period | Post-treatment period | atment<br>od |
|---|---|---|---|---|
| monitoring procedures to be applied to the patients apart from those of routine clinical practice) | Visit 1 | EoT (on-treatment visits) | Safety<br>Follow-up<br>visit | SVR12<br>Follow-up<br>visit |
| Written patient authorization form | X | | | |
| Inclusion/Exclusion Criteria | X | | | |
| Demographic information | X | | | |
| IL28B | X | | | |
| Relevant CHC disease characteristics | X | | | |
| Liver fibrosis stage | X | | | |
| CHC treatment history | X | | | |
| HCV genotype and subtype | X | | | |
| HCV RNA samples | X | X | | X |
| Clinical chemistry and hematology | X | X | | X |
| ABBVIE REGIMEN initiation documentation | X | | | |
| ABBVIE REGIMEN adherence | X | X | | |
| Concomitant medication | X | X | | X |
| Relevant medical history, co-morbidities | X | | | |
| SAE, non-serious AE and pregnancy reporting | × | × | × | × |

Time windows for reported clinical laboratory test results are described in the table 4.2

Table 4.2 – Analysis time windows

| Time point | Time Window |
|---|---|
| Visit 1 | Last value prior to start of study treatment (i.e. \( \le \) study day 1) |
| $EoT^1$ | Study day of last dose (from study day 56 to study day 98) |
| SVR12 | last value between 57 and 112 days post the study day of last dose |

presented in this case even if EoT \(\leq \)study day 55 (less than 8 weeks). The EoT time window will not be used for the target population analyses, actual collected EoT visit will be



### 4.1 Sample size<sup>1</sup>

60 patients will be included in this descriptive study without any prior sample size calculation.

### 4.2 Randomization and blinding

procedures are not applicable. This study is observational with one treatment group. Randomization and blinding

### 4.3 Planned analyses

No analyses for DMC meetings and no interim analysis are planned in the study. The only final statistical analysis report will be performed for this study.

### S General considerations

stop day of assessments and events. Study Day will be calculated from the reference start date, and will be used to show start/

"X<del>X</del>" domain of the database). Reference start date is defined as the day of the start treatment ("EXSTDTC" variable from

If the date of the event is on or after the reference date then study day = (date of event - reference date) + 1.

If the date of the event is prior to the reference date then study day = (date of event - reference date) - 1.

Baseline is defined as the measurement taken on Visit 1.

## **Analysis populations**

conventions adjustment for EoT. fulfill the eligibility criteria. Patients who prematurely discontinue earlier than study day 55 will be used in analyses on the target population with actual EoT time point without windowing The target population (TP) - all patients with signed written Patient Authorization, who

patients will be included to the NCP). Patients with  $EoT \le study day 55$  (less than 8 weeks) will be excluded from the CP (these treatment combination recommended in the current local label for their disease characteristics. The core population (CP) - all patients of the TP, who have started and received the

REGIMEN The safety population (SP) - all patients who received at least one dose of the ABBVIE

local label. The non-core population (NCP) – patients not receiving the treatment recommended in the

one of the following criteria: The core population with sufficient follow-up data (CPSFU) – all CP patients, who fulfil

evaluable HCV RNA data within the SVR12 time window

<sup>1</sup> This section is based on the section 9.11 "Study Size" of clinical study Protocol.



- response achieved at the last measurement on-treatment or post-treatment); a HCV RNA value ≥50 IU/mL at the last measurement post-baseline (i.e. no virological
- reported in the eCRF but date and value of the corresponding HCV RNA test is to AE) or incomplete efficacy information (e.g. virologic failure such as relapse is measurement on the SVR12 visit due to reasons related to safety (e.g. dropped out due missing). RNA <50 IU/mL at the last measurement post-baseline, but no HCV RNA

perform an additional HCV RNA test on the SVR12 visit) will be excluded from this analysis. for reasons not related to safety or effectiveness (e.g. lost-to-follow-up or patient not willing to treatment measurement, but had no HCV RNA measurements within the SVR12 time window In this way, only patients who had virological response at their last on-treatment or post-

follow-up data (CPSFU). Figure 6.1 illustrates the rule of patient's allocation in the core population with sufficient



Figure 6.1 – The core population with sufficient follow-up data (CPSFU) allocation

## 7 Statistical considerations

## 7.1 Standard descriptive statistics

minimum and maximum values. In quantitative tests the values less than LLoQ will be replaced to subjects with no missing data), mean, median, standard deviation (SD), interquartile range (IQR), 1/2 of LLoQ, the values more than ULoQ will be replaced to ULoQ. The data of continuous type will be presented with following statistics: n (the number of

percentages by categories will be based on the number of subjects with no missing data. number of subjects with no missing data), frequencies and percentages. Unless otherwise specified, The data of categorical type (including clinical evaluations) will be presented with n (the



following rules: The number of decimals for each descriptive statistical value will be determined by the

- mean, median and IQR: +1 decimal symbol compared to the analyzed variable values;
- standard deviation: +2 decimal symbols compared to the analyzed variable values;
- minimum and maximum values: the same as for the analyzed variable values;
- percentages will be rounded to one decimal symbol;
- confidence intervals will be presented with accuracy of the estimated value

## 7.2 Statistical tests and common calculations

The following arrangements will be applied:

- all tests will be two-sided with the default significant level 5%;
- confidence intervals will be 95% and will be determined using the Clopper-Pearson
- type I error values (p-values) will be rounded to four decimal symbols

calculated as (measurement at visit X – measurement at baseline). For quantitative measurements of clinical laboratory data, changes from baseline will be

## 7.3 Missing data

following rules will be used for the classification of AEs for AEs of the study period and AEs, which occurred before the start of treatment: If the information about adverse event start date and time is missing or incomplete, the

Table 7.1 – AEs missing management.

| is n | is k | is n | is k | is n | is n | |
|---|---|---|---|---|---|---|
| is missing | is known | is missing | is known | is missing | is missing | Day |
| is missing | is missing | is known | is missing | is missing | is known | Month |
| is missing | is missing | is missing | is known | is known | is known | Year |
| | AE will be classified as AE of the study period | | administration date | AE will be classified as AE of the study period, | AE will be classified as AE of the study period, if month and year ≥ month and year of the first study drug administration date | Processing |

## 7.4 Multicenter studies

Data from all centers will be merged and analyzed as one population for all study endpoints The study will take place in 5-7 centers (national and regional hospitals/outpatient services).

## 7.5 Multiple comparisons

No adjustments for multiplicity are required

## Summary of study data



Each study variable will be analyzed for relevant population.

and study period/assessment (i.e. time point), where applicable. Unless otherwise specified all raw data will be listed and sorted by unique subject identifier

prior and concurrent medications will be reported for the core population (CP). Demographic and baseline characteristics, concurrent illnesses and medical conditions,

subtype, fibrosis status and treatment experienced or naīve. The results will be presented overall and for the CP analysis groups based on genotype

CP analysis groups by the following parameters: According to the eligibility criteria of this study<sup>1</sup>, only patients with genotype 1b and Child Pugh A cirrhosis will be included in this study. In this way, the results will be presented for the

- cirrhosis score<sup>2</sup> (5 or 6);
- treatment experienced or naīve patients<sup>3</sup> (with/without prior treatment for CHC).

the safety population (SP) overall only (without the CP analysis grouping). conditions, prior and concurrent medications will be reported for the target population (TP) and Additionally demographic and baseline characteristics, concurrent illnesses and medical

## Subject disposition

written patient authorization form and will include the following results: Subject disposition will be represented in tables and listings for all patients who signed the

- the number of subjects who signed the written patient authorization form:
- the number of subjects in each analyzed population;
- the number of subjects who has HCV RNA assessment on SVR12;
- the number of subjects without HCV RNA assessment on SVR12 and the reasons for it;
- corresponding violated inclusion/exclusion criteria. number of patients with the violations of the eligibility criteria and the

### 8.2 **Protocol deviations**

The presentation of Protocol deviations is not planned in this study

## Demographic and baseline variables

following parameters, which are evaluated on visit 1: Tables with descriptive statistics in accordance with section 7.1 will be presented for the

- demographics and anthropometric characteristics:
- gender;
- race/ethnic origin
- height;
- weight;
- BMI [weight (kg) / height (m<sup>2</sup>)];
- duration of HCV infection diagnosis (in years);
- IL28B genotypes;

Sections 9.6 "Inclusion Criteria" and 9.7 "Exclusion Criteria" of the clinical study Protocol

 Data MATRIX Ltd.

Parameter "CIRRHOSIS SCORE" from eCRF form "CHC DISEASE CHARACTERISTICS".

Parameter "Prior treatment for CHC" from eCRF form "MOST RECENT PRIOR THERAPY FOR CHC"



- most likely mode of HCV infection;
- liver biopsy results (staging by histopathological scoring system):
- elastography (kPa);
- FibroTest;
- presence of esophageal varices;
- history of liver decompensation;
- Child Pugh score;
- alcohol consumption:
- alcohol use;
- number of units/drinks per week (for patients who regular use alcohol).

All corresponding listings will be presented.

## 8.4 Concurrent illnesses and medical conditions

LLC SOP [3] and will be presented in listings and tables. summarized by system organ class (SOC) and preferred term (PT) according Data MATRIX Medical history will be coded using the MedDRA version 20.0 (or further updating) and

following parameters, which are evaluated on visit 1: Tables with descriptive statistics in accordance with section 7.1 will be presented for the

- co-infection information:
- presence of co-infection with other relevant diseases;
- CD4 T-cell count (for HIV co-infected patients);
- HIV-RNA test results (for HIV co-infected patients);
- liver and/or CHC related co-morbidities;
- other co-morbidities.

## 8.5 Prior and concurrent medications

medications will be presented in a separate listings and tables. time of the study completion) according Data MATRIX LLC SOP [3]. Prior and concurrent All medications will be coded using WHODD version Jun 2015 (or actual version on the

determined using "CO-MEDICATION" flag in the CMCAT variable of CM domain of the database. in the CMCAT variable of CM domain of the database. Concurrent medications will be Prior medication will be determined using "MOST RECENT PRIOR THERAPY FOR CHC"

Additionally listings will contain the following information for prior CHC therapy:

- presence of prior treatment for CHC;
- generic drug name;
- initial dose (by generic drug name groups and units groups);
- start frequency (by generic drug name groups);
- duration (by generic drug name groups, in weeks);
- outcome prior treatment.

## 9 Effectiveness analysis

with separate tables for each population as the result. Tables for equal sets (contain exactly the All analyses of effectiveness will be performed on the TP, CP and CPSFU populations



only. same patients) will not be presented, equal sets will be pointed in the footnote with description

The following effectiveness outcomes will be included in the analyses:

- SVR12 achieving;
- virological response at EoT;
- patients with at least one and each of SVR12 non-response categories:
- relapse during treatment phase;
- relapse after EoT;
- failure to suppress;
- premature study drug discontinuation with no on-treatment virologic failure;
- missing SVR12 data.

analyzed with the following definitions: detection higher than 50 IU/mL and may vary across laboratories, effectiveness outcomes will be Due to the fact that in the Russian clinical practice tests for HCV RNA often have limit of

- SVR12 achieving (single last HCV RNA value <50 IU/mL or undetectable/negative 12 weeks after the last actual dose of the ABBVIE REGIMEN);
- virological response (HCV RNA <50 IU/mL or undetectable/negative) at EoT;
- patients with at least one and each of SVR12 non-response categories:
- relapse during treatment phase (breakthrough, i.e. at least one documented HCV IU/mL or positive during treatment); RNA value <50 IU/mL or undetectable/negative followed by HCV RNA value ≥50
- the last on-treatment HCV RNA measurement followed by HCV RNA ≥50 IU/mL or relapse after EoT (HCV RNA value <50 IU/mL or undetectable/negative at EoT or at positive post-treatment);
- failure to suppress (each measured on-treatment HCV RNA value >50 IU/mL
- premature study drug discontinuation with no on-treatment virologic failure
- missing SVR12 data and/or none of the above criteria.

categories. Figure 9.1 illustrates the patient's distribution by SVR12 response/non-response





Figure 9.1 – Patient's distribution by SVR12 response/non-response categories

will be repeated for patients in subgroup without missing SVR12 data category. effectiveness outcomes and will be presented according the section 7.1. Also frequency tables Frequencies and percentages with 95% confidence intervals will be calculated for each

groups, since not each covariate might be predictive in each patient group. of exploratory nature, data driven, and will be repeatedly performed for various CP analysis EoT) will be analyzed using univariate logistic regression, if applicable. These analyses will be Effectiveness endpoints (SVR12 achieving, virological response at EoT and relapse after

(fixed effect or covariate): The following parameters can be included in the univariate models as explanatory variables

- treatment experience (with/without prior treatment for CHC);
- Child Pugh score;
- result of FibroTest;
- history of liver decompensation;
- gender;
- race;

BMI;

- laboratory hematology<sup>1</sup>:
- hemoglobin;
- platelets;
- prothrombin time
- laboratory clinical chemistry:

smallest units groups the corresponding covariate will be deleted from the analysis. <sup>1</sup> Note that all Hematology variables and all Clinical Chemistry should be in the same units. If it is impossible to bring units to the same the smallest units groups will be accepted as missing. If it is impossible to identify the



- ASI
- Gamma-GT;
- total bilirubin;
- albumin;
- creatinine clearance;
- alpha-1-fetoprotein.

value < 0.25 in the corresponding univariate logistic regression analysis MLR (if applicable) which consider only covariates in the selection procedure with a p-Additionally, after univariate model analyses all effectiveness endpoints can be analyzed

using following SAS script: To avoid the multicollinearity problem all possible explanatory variables will be examined

ods graphics on;
PROC CORR data=<dataset> plots=all;
VAR <variables>;
RUN;
ods graphics off;

considered and managed. All solutions about an explanatory variables choosing will be of exploratory nature, data driven, and will be described with presenting of results of the "PROC" CORR" SAS procedure. Statistical significant correlated variables with correlation coefficient > 40 should be

0.05. A p-value <0.05 condition will be used for the covariates to stay in the model in a backward elimination step. procedure LOGISTIC with statement SELECTION = Backward selection procedures will be applied to generate the final MLR models esing the **BACKWARD** and **SLENTRY** 

Odds ratio with 95% Wild CI, p-values will be presented for each predictor

analyses endpoint). All data for effectiveness analyses will be listed in separate listings (for each effectiveness

### 10 Safety analysis

Safety analysis will be conducted on the safety population (SP).

The following parameters will be analyzed:

- study drug exposure;
- adverse events;
- pregnancies;
- clinical laboratory evaluations.

### 10.1 Exposure

following parameters: Tables with descriptive statistics in accordance with section 7.1 will be presented for the

actual duration ABBVIE REGIMEN (in days);

 Data MATRIX Ltd.

<sup>&</sup>lt;sup>1</sup> Note that MLR is possible ONLY if more than one explanatory variables will have a p-value <0.25 in the corresponding univariate logistic regression analysis.



## P16-253 (CITRIN) \_ STATISTICAL ANALYSIS PLAN \_ FINAL 2.0 \_ 16 Mar 2018

- the number of patients with collected deviating duration reasons;
- adherence Dasabuvir separately): ABBVIE REGIMEN (calculated for Paritaprevir/R-Ombitasvir and for
- percentage of target dose taken in treatment intervals (weeks 1-4, 5-8 and 9-12) for Paritaprevir/R-Ombitasvir and for Dasabuvir;
- percentage of patients who missed of study drug administration for at least 7 days in a row

All corresponding listings will be presented.

## 0.2 Adverse events

Only treatment-emergent adverse events will be analyzed.

initiation of study drug through 30 days post-study drug dosing. Treatment-emergent AE is any reported event that begins or worsens in severity after

tabulated in the report with grouping by primary system organ class (SOC) and preferred term (PT). All analyzed AEs will be coded using the MedDRA version 20.0 (or further updating) and

with this AE emergence as well as the total number of episodes this AE for a diagnosis. The frequency of a specific AE occurrence will be presented by the proportion of patients

presented: The following tables with descriptive statistics in accordance with section 7.1 will be

- all AE / SAE;
- AE / SAE by severity;
- AE / SAE by relationship to the study drug.

(relationship to the study drug) in each SOC and each PT level as well as Total level. be considered. At the same time, each patient will be counted only once with highest severity (relationship to the drug) in each patient, while in the Total category all AEs of this patient will following rules. Each SOC / PT category will include only the AEs with the highest severity Tables of AE/SAE by severity (relationship to the study drug) will be prepared using the

errors will be provided. Also all AEs will be presented in listings. Additional listings for unintended medication

### 10.3 Pregnancies

and pregnancies episodes will be reported in the listing Female subjects will be tested for pregnancy at each study visit. The results of these tests

## 10.4 Clinical laboratory evaluations

Clinical laboratory evaluations include the following parameters:

- hematology results;
- blood chemistry results.

tables and presented in listings: The following parameters, which are evaluated at each study visit, will be analyzed in

- hematology:
- hemoglobin;
- platelets;
- prothrombin time (seconds);



- prothrombin time (INR);
- blood chemistry:
- ALT;
- AST;
- GGT;
- total bilirubin;
- alpha-1-fetoprotein;
- albumin;
- creatinine;
- creatinine clearance.

accordance with section 7.1 as the following outputs: The results of clinical laboratory evaluations statistical analysis will be represented in

- tables with descriptive statistics of measurement values and changes from baseline (visit 1);
- frequency tables of out of range and clinically significant evaluates will be presented;
- shift tables based on clinical evaluation of measurements at visit 1.

## 10.5 Other safety measures

No other safety measures will be analysed in this study.



### P16-253 (CITRIN) STATISTICAL ANALYSIS PLAN FINAL 2.0 16 Mar 2018

## 11 Pharmacokinetics

No pharmacokinetic and pharmacodynamic parameters will be analyzed in this study.

### 12 Other analyses

No other analyses will be performed in this study.

## 13 Interim analyses and data monitoring

No interim analysis is planned for this study.

## 14 Technical details and reporting conventions

and listings in English. database lock. The results of statistical analysis will be presented in the form of tables, figures will be prepared in the Microsoft Office Word (.docx) format after the end of data collection and Statistical analysis will be performed using SAS 9.4. One (final) statistical analysis report

## 15 Summary of changes to the Protocol

This SAP is fully consistent with the clinical study Protocol.

### 16 List of TFLs

### 16.1 Tables

## Subjects Disposition

```
Table 1.1 - Subjects Dispositions
Table 1.2 - The reasons of early wirthdrawal
Table 1.3 - Violation of eligibility criteria
```

## Demographics and anthropometric characteristics

```
Table Table
                            Table
                                                      Table
                                                                   Table
                                                                                Table
                                          [CP]
                                                                1.4.1 -
1.4.4
1.4.5
1.4.6
                                                     1.4.
                                                       ω
    1 1
                                                                  Demographics and anthropometric characteristics (prior
Demographics and Demographics and
                            Demographics and anthropometric characteristics (Child Pugh
                                                                                Demographics and anthropometric characteristics
                                                     Demographics
                                                     and anthropometric
 anthropometric anthropometric
 characteristics characteristics
                                                      characteristics
 [TP]
                                                                                [CP]
                                                     (treatment-experienced
                                                                   treatment
                          score groups) [CP]
                                                                  groups)
```

## CHC disease characteristics

```
Table
                                 Table
1.5.5.
5.5.4
6.5.5
                              1.5.1
CHC
                               CHC
                                                      CHC
         C disease characteristics C disease characteristics C disease characteristics C disease characteristics
 disease characteristics
                                                      disease
                                                      characteristics
(Child Pugh score groups) [CP] [TP] [SP]
                               (prior treatment groups) [CP]
(treatment-experienced groups)
                                 [CP]
```

### Liver fibrosis stage

```
Table
                                Table
                          Table
                                          Table
                        1.6.1
1.6.2
1.6.3
11.
6.6.
6.4
                        Liver
Liver
Liver
        Liver
Liver
 Liver
                         fibrosis
fibrosis
 fibrosis
         fibrosis
                 fibrosis
                                          fibrosis
               stage
stage
stage
stage
         stage
(prior treatment groups) [CP]
(treatment-experienced groups)
(Child Pugh score groups) [CP]
[TP]
[SP]
```



### P16-253 (CITRIN) STATISTICAL ANALYSIS PLAN EZ A 2.0 16 Mar 2018

```
Table
                             Table
               Table
                                            Table
                                                                                         Alcohol consumption
1.7.3 - Alcohol consumption
1.7.4 - Alcohol consumption
1.7.5 - Alcohol consumption
1.7.6 - Alcohol consumption
                                                       1.7.2
                                                         Alcohol
                                                                         Alc
                                                                         cohol
                                                          consumption
                                                                      consumption
              (Child Pugh
 [SP]
                                                                      [CP]
                            (prior treatment groups) [CP] (treatment-experienced groups) [CP] (Child Pugh score groups) [CP]
```

## Liver and/or CHC related co-morbidities

```
Table
Table
                   Table
                              Table
                                         Table
                                                 Table
1.8.8.3
1.8.3
                                       1.8.1
  1 1 1
                                        Liver
Liver
Liver and/or CHC related
Liver and/or CHC related
Liver and/or CHC related
Liver and/or CHC related
                                        and/or and/or
                                        CHC
                                       related
d co-morbidities
d co-morbidities
co-morbidities
                              co-morbidities
                                        co-morbidities co-morbidities
[SP]
                   (prior treatment groups) [CP]
(treatment-experienced groups)
(Child Pugh score groups) [CP]
                                        (prior treatment
                              [CP]
```

## Other co-morbidities

```
Table
                    Table
                             Table
                                       Table
                                                 Table
11111
  1 1 1
Other co-morbidities
Other co-morbidities
Other co-morbidities
Other co-morbidities
Other co-morbidities
                                                Other
                                                co-morbidities
(treatment-experienced groups)
(Child Pugh score groups) [CP]
[TP]
                                                [CP]
                                      (prior
                                      treatment groups) [CP]
                              [CP]
```

### Co-infections

```
Table
                       Table
                                              Table
  Table
                                    Table
1.10.3 -
1.10.4 -
1.10.5 -
1.10.6 -
                                 1.10.1
            Co-infections
Co-infections
                                  Co-infections
Co-infections
 Co-infections
                                                         Co-infections
s [CP]
s (prior treatment groups) [CP]
s (treatment-experienced groups) [
s (Child Pugh score groups) [CP]
s [TP]
s [SP]
```

### VIH most recent test results

```
Table Table
                Table
                         Table
                                Table
                                        Table
1.111.3
 HIV most
HIV most
HIV most
                                HIV most
most
recent test
recent test
recent test
recent test
recent test
                                       recent
                                       test
 results results results
                               results results
s [CP]
s (prior treatment groups) [CP]
s (treatment-experienced groups)
s (Child Pugh score groups) [CP]
s [TP]
s [SP]
                         [CP]
```

### Prior Medications for CHC

```
Table
                 Table
                        Table
                                 Table
                                        Table
1.112.1
Prior Medications
Prior Medications
Prior Medications
                                Prior Medications
Prior Medications
                        Prior Medications
 for
for
                       for
for
                                        for
 CHC
CHC
CHC
CHC
(treatment-experienced groups)
(Child Pugh score groups) [CP]
[TP]
                                        [CP]
                              (prior treatment groups) [CP]
                        [CP]
```

## Concurrent Medications for CHC

```
Table
                                                      Table
1.113.
1.113.
1.113.
1.113.
1.113.
1.113.
1.113.
1.113.
          Concurrent Medications
Concurrent Medications
  Concurrent
                                Concurrent
                                         Concurrent
                                                     Concurrent
                               Medications
Medications
  Medications
                                                     Medications
 H, H, H, H, H, H, O O O O O O O O O
 CHC
CHC
CHC
CHC
C [CP]
C (prior treatment groups) [CP]
C (treatment-experienced groups)
C (Child Pugh score groups) [CP]
C [TP]
C [SP]
                                 [CP]
```

### Effectiveness analysis 1 1

Table Table

2.1.1.1 2.1.1.2

Percentage fPercentage

for

for

effectiveness e

endpoints

[TP]

endpoints

ļ,

subgroup

without

missing

SVR12

data

```
Table
                                                                                                                                                                                             Table
                                                                                                                                                                                                                                                        Table
1 \quad 1 \quad 1 \quad 1 \quad 1 \quad 1
                                                                                                                                                                                        SVR12 achieving. Univa
SVR12 achieving. Multi
Virological response at
     Relapse
                                                                    Relapse
                                                                                                                         Virological
                          achieving. Univariate logistic regression results [TP] achieving. Multiple logistic regression results [gical response at EoT. Univariate logistic regressions results [action regression results [action regressions results [action regressions results [action regressions results [action results [action regressions results [action regressions results [action regressions results [action regressions results [action results [action regressions results [action regressions results [action regressions results [action regressions results [action regressions results [action regression regression regress
     after
     EOT.
     Multiple
logistic
logistic
     regression
     [TP]
                                                                                                                                                                                                   [TP]
```



## P16-253 (CITRIN) STATISTICAL ANALYSIS PLAN FINAL 2.0 16 Mar 2018

```
Table Table
                                                               Table
Table
                                                                                                                                                                                                                                                          Table
                                                                                                                                                                                                                                                                                Table
                                                                                                                                                                                                                                                                                                      Table
                                                                                                                                                                                                                                                                                                                                                                                                                                               Table
                                                                                                                                                                                   Table 2.3.1.1
Table 2.3.1.2
                                                                                                                                                                                                                                                                                                                                                                                                                            [CP]
                                            Table
                                                                                                                                                                  [CPSFU]
                                                                                                                                                                                                                                                                                                                             Table
2.2.1.1
                                                                                                                                                                                                                                                                                                                                                                                                                                               2.2.1.2
                                                                                                                                                                                                           ı
      1 1
                                                                                                                                                                                                                                                                 1 1 1
                                                                                                                                                                                                         Percentage for effectiveness endpoints [CPSFU]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                   Percentage for effectiveness endpoints
                                                                                                                                                                                                                                                    SVR12 achieving. Univariate logistic regression results [TP] SVR12 achieving. Multiple logistic regression results [TP] Virological response at EoT. Univariate logistic regressions results [Virological response at EoT. Multiple logistic regression respense after EoT. Univariate logistic regressions results [TP] Relapse after EoT. Multiple logistic regression results [TP]
Virological response at EoT. Multiple logistic regression Relapse after EoT. Univariate logistic regressions results [C] Relapse after EoT. Multiple logistic regression results [A]
                                                              SVR12 achieving. Univariate logistic regression results [CPSFU] SVR12 achieving. Multiple logistic regression results [CPSFU] Virological response at EoT. Univariate logistic regressions results
                                                                                                                                                                                                                                                                                                                                                                                                                                               Percentage
                                                                                                                                                                                   Percentage for effectiveness endpoints in
                                                                                                                                                                                                                                                                                              achieving. Univariate logistic regression results [TP] achieving. Multiple logistic regression results [TP] sgical response at EoT. Univariate logistic regressions results ogical response at EoT. Multiple logistic regression result
                                                                                                                                                                                                                                                                                                                                                                                                                                               for effectiveness endpoints
                                                                                                                                                                                                                                                                                                                                                                                                                                                                     [CP]
                  regressions results [CPSFU]
                                                                                                                                                                                                                                                                                                                                                                                                                                             in subgroup without missing
                                                                                                                                                                                   subgroup without missing
     [CPSFU]
                                              results
                                                                                                                                                                                                                                                                                                     results
                                                                                                                                                                                                                                                                                                      [TP]
s [TP]
                                                                                                                                                                                     SVR12
                                                                                                                                                                                                                                                                                                                                                                                                                                                SVR12 data
                                              [CPSFU]
                                                                                                                                                                                     data
```

### Exposure

Table AbbVie REGIMEN intake

### events

```
Table
                   Table
                             Table
Adverse
Serious
                  Adverse
Serious
                                    Adverse
Serious
  adverse
                   adverse events by relationship to the study drug
                           events by relationship to the study drug
          events
                                     adverse events
                                              events
           by severity
  events by
  severity
```

### Hematology

```
Table 3.3.1 -
Table 3.3.2 -
Table 3.3.3 -
   Hematology.Hematology.Hematology.
 Descriptive statisti
Clinical assessments
Shift table
                                statistics
```

### Blood chemistry

```
Table 3.4.1 - Blood
Table 3.4.2 - Blood
Table 3.4.3 - Blood
chemistry.
chemistry.
chemistry.
Descriptive
Clinical ass
Shift table
                 assessments
                             statistics
```

### 16.2 **Figures**

No figures are planned in the study.

### 16.3 Listings

## Patients disposition

```
Listing 1.1 - Disposition: analysis populations
Listing 1.2 - Disposition: subject visits
Listing 1.3 - Disposition: study completion
Listing 1.4 - Violation of inclusion/exclusion criteria
```

## Demographics and baseline characteristics

```
Listing
Listing
                                                                                                    Listing
                                                                                                                                                                               Listing
                                                                         Listing
                                                                                                                             Listing
                                                                                                                                                        Listing
ing 2.1 - Demographics and anthropometric charactering 2.2 - CHC disease characteristics

Ing 2.3.1 - Patients co-infections

Ing 2.3.2 - HIV co-infection

Ing 2.4 - Medical History: Other Co-Morbidities

Ing 2.5 - Medical History: liver and/or CHC relate

Ing 2.6.1 - Most Recent Prior Therapy For CHC

Ing 2.6.2 - Co-medication

Ing 2.7.1 - Alcohol consumption

Ing 2.7.2 - Patients with regular alcohol consumpt
    alcohol consumption
                                                                                                                                                                                                                                       characteristics
                                                                                                          related co-morbidities
```



## P16-253 (CITRIN) \_ STATISTICAL ANALYSIS PLAN FINAL 2.0 \_16 Mar 2018

Listing 2.8 - Interleukin 28B genotypes

## Effectiveness analysis Listing 3.1 - HCV RNA

### Safety analysis

Listing 4.1 - Adverse Events
Listing 4.2.1 - ABBVIE REGIMEN: exposure
Listing 4.2.2 - ABBVIE REGIMEN: adherence
Listing 4.3 - Pregnancy
Listing 4.4 - Hematology results
Listing 4.5.1 - Blood chemistry results
Listing 4.5.2 - Optional blood chemistry results

### 17 References

- 1) Committee for Proprietary Medicinal Products (CPMP). International Conference on Harmonisation (ICH) Topic E9: Note for Guidance on Statistical Principles for Clinical Trials; September 1998.
- DataMatrix\_SOP\_STAT001\_Statistical Principles\_ver.2.0\_June 2016.
   DataMatrix\_SOP\_DM010\_Dictionary Management and Data Coding\_ver.2.0\_August



### 18 Tables shells

### **Subjects disposition**

AbbVie LLC P16-253 (CITRIN)

### Table 1.1 Subjects Disposition

All patients Page X of X

| | Total<br>n (%) |
|------------------------------------------------------------|----------------|
| Subjects who signed the written patient authorization form | XX |
| The target population (TP) | XX (XX.X) |
| The core population (TP) | XX (XX.X) |
| The safety population (SP) | XX (XX.X) |
| The non-core population (NCP) | XX (XX.X) |
| The core population with sufficient follow-up data (CPSFU) | XX (XX.X) |

n: the number of subjects within a specific category.

Percentages were calculated from the number of subjects who signed the written patient authorization form.



AbbVie LLC P16-253 (CITRIN)

### Table 1.2 The reasons of early withdrawal

The target population Page X of X

| | Total |
|-------------------------------------------------|-----------|
| | (N = XX) |
| | n (%) |
| Subjects with HCV RNA assessment on SVR12 | XX (XX.X) |
| Subjects without HCV RNA assessment on SVR12 | XX (XX.X) |
| Reason if HCV RNA assessment on SVR12 not done: | |
| Failure to return | XX (XX.X) |
| Insufficient virological response | XX (XX.X) |
| Withdrawn consent | XX (XX.X) |
| Death | XX (XX.X) |
| • • • | ••• |

N: the number of subjects in the target population. n: the number of subjects within a specific category. Percentages were calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.3 Violation of eligibility criteria

The target population Page X of X

| | Total |
|---|---|
| | (N = XX) |
| | n (%) |
| Patients with violation of inclusion criteria | XX (XX.X) |
| Inclusion criterion #1 | XX (XX.X) |
| Inclusion criterion #2 | XX (XX.X) |
| ••• | • • • |
| Patients with violation of exclusion criteria | XX (XX.X) |
| Exclusion criterion #1 | XX (XX.X) |
| Exclusion criterion #2 | XX (XX.X) |
| ••• | • • • |
| Subject has fulfilled all the inclusion and does not meet any exclusion criteria and is eligible for the trial | XX (XX.X) |

N: the number of subjects in the target population. n: the number of subjects within a specific category. Percentages are calculated as (100 x n/N).



### Demographic and anthropometric characteristics

AbbVie LLC P16-253 (CITRIN)

### Table 1.4.1 Demographics and anthropometric characteristics

The core population Page X of X

| | | Total |
|---------------------------------|-------|-----------|
| | | (N=XX) |
| Age (years) | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| IQR | | XX.X |
| Min | | XX |
| Max | | XX |
| Gender | | |
| n | | XX |
| Male | n (%) | XX (XX.X) |
| Female | n (%) | XX (XX.X) |
| Race | | |
| n | | XX |
| White/Caucasian | n (%) | XX (XX.X) |
| Black | n (%) | XX (XX.X) |
| Asian/Oriental | n (%) | XX (XX.X) |
| Native American/American Indian | n (%) | XX (XX.X) |
| Other | n (%) | XX (XX.X) |
| Weight (kg) | | |
| ••• | | • • • |
| Height (cm) | | |
| ••• | | • • • |
| BMI (kg/m^2) | | |
| • • • | | |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ . IQR: interquartile range. Body Mass Index (BMI): weight (kg) / [height (m)^2]. Age is calculated as the number of full years between the date of birth and the date of signing the written patient authorization form.



AbbVie LLC P16-253 (CITRIN)

### Table 1.4.2 Demographics and anthropometric characteristics (prior treatment groups)

The core population Page X of X

| | | Treatment-<br>experienced<br>(N=XX) | Naïve<br>(N=XX) |
|--------------|-------|-------------------------------------|-----------------|
| Age (years) | | | |
| | | | • • • |
| Gender | | | |
| • • • | • • • | • • • | • • • |
| Race | | | |
| • • • | | • • • | • • • |
| Weight (kg) | | | |
| ••• | | | • • • |
| Height (cm) | | | |
| | | • • • | • • • |
| BMI (kg/m^2) | | | |

N: the number of subjects in the prior treatment groups of the core population. n: the number of valid measurements. IQR: interquartile range. Body Mass Index (BMI): weight (kg) / [height (m)^2]. Percentages are calculated as  $(100 \times n/N)$ . Age is calculated as the number of full years between the date of birth and the date of signing the written patient authorization form.



AbbVie LLC P16-253 (CITRIN)

### Table 1.4.3 Demographics and anthropometric characteristics (treatment-experienced groups)

The core population Page X of X

| | | PEG-INF alpha (N=XX) | non-PEG-INF<br>alpha<br>(N=XX) | INF all (N=XX) | Ribavirin<br>(N=XX) |
|---|---|---|---|---|---|
| Age (years) | | | | | |
| • • • | | • • • | • • • | • • • | • • • |
| Gender | | | | | |
| • • • | • • • | • • • | • • • | • • • | • • • |
| Race | | | | | |
| • • • | | | • • • | | • • • |
| Weight (kg) | | | | | |
| ••• | | | • • • | | |
| Height (cm) | | | | | |
| ••• | | • • • | | | |
| BMI (kg/m^2) | | | | | |
| | | • • • | | • • • | |

N: the number of subjects in the treatment-experienced groups of the core population. n: the number of valid measurements. IQR: interquartile range. Body Mass Index (BMI): weight (kg) / [height (m)^2]. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated). Age is calculated as the number of full years between the date of birth and the date of signing the written patient authorization form.



AbbVie LLC P16-253 (CITRIN)

Table 1.4.4 Demographics and anthropometric characteristics (Child Pugh score groups)

The core population

he core population Page X of X

| | | Score 5 (N=XX) | Score 6 (N=XX) |
|--------------|-----|----------------|----------------|
| Age (years) | | | |
| • • • | | | • • • |
| Gender | | | |
| • • • | ••• | • • • | • • • |
| Race | | | |
| • • • | ••• | • • • | • • • |
| Weight (kg) | | | |
| ••• | | • • • | • • • |
| Height (cm) | | | |
| ••• | | | |
| BMI (kg/m^2) | | | |
| ••• | | | |

N: the number of subjects in the Child Pugh score groups of the core population. n: the number of valid measurements. IQR: interquartile range. Body Mass Index (BMI): weight (kg) / [height (m)^2]. Percentages are calculated as (100 x n/N). Age is calculated as the number of full years between the date of birth and the date of signing the written patient authorization form.

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.4.1, tables for the target and the safety populations will be constructed:

Table 1.4.5 Demographics and anthropometric characteristics Table 1.4.6 Demographics and anthropometric characteristics



### **CHC** disease characteristics

AbbVie LLC P16-253 (CITRIN)

### Table 1.5.1 CHC disease characteristics

The core population Page X of X

| | | Total<br>(N=XX) |
|------------------------------------------------|-------|-----------------|
| Duration of HCV infection diagnosis (in years) | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| IQR | | XX.X |
| Min | | XX |
| Max | | XX |
| Most likely mode of HCV infection | | |
| n | | XX |
| Blood transfusions | n (%) | XX (XX.X) |
| Dental procedures | n (%) | XX (XX.X) |
| | | • • • |
| IL28B genotypes | | |
| rs12979860 | | |
| n | | XX |
| CC | n (%) | XX (XX.X) |
| CT | n (%) | XX (XX.X) |
| TT | n (%) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) |
| rs8099917 | | |
| n | | XX |
| GG | n (%) | XX (XX.X) |
| TG | n (%) | XX (XX.X) |
| TT | n (%) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC

### P16-253 (CITRIN)

### Table 1.5.2 CHC disease characteristics (prior treatment groups)

The core population Page X of X

| | | Treatment-<br>experienced<br>(N=XX) | Naïve<br>(N=XX) |
|---|---|---|---|
| Duration of HCV infection diagnosis (in years) | | | |
| ••• | | • • • | • • • |
| Most likely mode of HCV infection | | | |
| ••• | • • • | • • • | • • • |
| IL28B genotypes rs12979860 | | | |
| ••• | • • • | • • • | • • • |
| rs8099917 | | | |
| ••• | | ••• | |

N: the number of subjects in the prior treatment groups of the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.5.3 CHC disease characteristics (treatment-experienced groups)

The core population Page X of X

| | | PEG-INF alpha (N=XX) | non-PEG-INF alpha<br>(N=XX) | INF all (N=XX) | Ribavirin<br>(N=XX) |
|---|---|---|---|---|---|
| Duration of HCV infection diagnosis (in years) | | | | | |
| ••• | | • • • | ••• | • • • | • • • |
| Most likely mode of HCV infection | | | | | |
| ••• | • • • | • • • | ••• | • • • | • • • |
| IL28B genotypes rs12979860 | | | | | |
| rs8099917 | | | | | |
| ••• | | | | | |

N: the number of subjects in the prior treatment groups of the core population. n: the number of valid measurements. Percentages are calculated as (100 x n/N).

PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).



AbbVie LLC P16-253 (CITRIN)

### Table 1.5.4 CHC disease characteristics (Child Pugh score groups)

The core population Page X of X

| | | Score 5 (N=XX) | Score 6<br>(N=XX) |
|---|---|---|---|
| Duration of HCV infection diagnosis (in years) | | | |
| ••• | | • • • | • • • |
| Most likely mode of HCV infection | | | |
| ••• | • • • | • • • | • • • |
| IL28B genotypes rs12979860 | | | |
| ••• | • • • | • • • | • • • |
| rs8099917 | | | |
| ••• | | | |

N: the number of subjects in the prior treatment groups of the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.5.1, tables for the target and the safety populations will be constructed:

Table 1.5.5 CHC disease characteristics Table 1.5.6 CHC disease characteristics



### Liver fibrosis stage

AbbVie LLC P16-253 (CITRIN)

### Table 1.6.1 Liver fibrosis stage

The core population Page X of X

| | | Total |
|---------------------------------------------|------|-------------|
| | , | N=XX) |
| | r | n (%) |
| Staging by histopathological scoring system | | |
| Elastography (kPa) | | |
| n | | XX |
| <8.8 | XX | (XX.X) |
| 8.8-<9.6 | XX | (XX.X) |
| 9.6-<14.6 | XX | (XX.X) |
| >=14.6 | XX | (XX.X) |
| FibroTest | | |
| n | | XX |
| <=0.21 | XX | (XX.X) |
| 0.22-0.27 | XX | (XX.X) |
| 0.28-0.31 | | (XX.X) |
| ••• | | ••• |
| Presence of esophageal varices | | |
| n | | XX |
| Yes | XX | (XX.X) |
| No | | (XX.X) |
| Unknown | | (XX.X) |
| History of liver decompensation | | |
| n | | XX |
| No, never decompensated | XX | (XX.X) |
| Yes, but currently compensated | | (XX.X) |
| res, suc currencry compensaced | 2121 | (2121 • 21) |
| Child Pugh score | | |
| n | | XX |
| 5 | XX | (XX.X) |
| 6 | XX | (XX.X) |
| • • • | | |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as (100 x n/N).



AbbVie LLC P16-253 (CITRIN)

### Table 1.6.2 Liver fibrosis stage (prior treatment groups)

The core population Page X of X

| | Treatment-<br>experienced<br>(N=XX)<br>n (%) | Naïve<br>(N=XX)<br>n (%) |
|---|---|---|
| Staging by histopathological scoring system Elastography (kPa) | | |
| ••• | • • • | |
| FibroTest | | |
| ••• | • • • | • • • |
| Presence of esophageal varices | | |
| ••• | • • • | • • • |
| History of liver decompensation | | |
| ••• | • • • | • • • |
| Child Pugh score | | |
| ••• | | |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.6.3 Liver fibrosis stage (treatment-experienced groups)

The core population Page X of X

| | PEG-INF alpha<br>(N=XX)<br>n (%) | non-PEG-INF alpha<br>(N=XX)<br>n (%) | INF all (N=XX) n (%) | Ribavirin<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| Staging by histopathological scoring system Elastography (kPa) | | | | |
| ••• | • • • | • • • | • • • | • • • |
| FibroTest | | | | |
| ••• | • • • | • • • | • • • | • • • |
| Presence of esophageal varices | | | | |
| • • • | • • • | • • • | • • • | • • • |
| History of liver decompensation | | | | |
| ••• | • • • | ••• | • • • | • • • |
| Child Pugh score | | | | |
| ••• | | | | |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).



AbbVie LLC P16-253 (CITRIN)

### Table 1.6.4 Liver fibrosis stage (Child Pugh score groups)

The core population Page X of X

| | Score 5<br>(N=XX)<br>n (%) | Score 6<br>(N=XX)<br>n (%) |
|---|---|---|
| Staging by histopathological scoring system Elastography (kPa) | | |
| ••• | • • • | |
| FibroTest | | |
| ••• | • • • | • • • |
| Presence of esophageal varices | | |
| ••• | ••• | • • • |
| History of liver decompensation | | |
| • • • | | |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.6.1, tables for the target and the safety populations will be constructed:

Table 1.6.5 Liver fibrosis stage Table 1.6.6 Liver fibrosis stage


### **Alcohol consumption**

AbbVie LLC P16-253 (CITRIN)

### Table 1.7.1 Alcohol consumption

The core population Page X of X

| | | Total |
|---------------------------------|-------|-----------|
| | | (N=XX) |
| Alcohol use | | |
| n | | XX |
| Ex-drinker | n (%) | XX (XX.X) |
| None | n (%) | XX (XX.X) |
| Yes, occasional | n (%) | XX (XX.X) |
| Yes, regular | n (%) | XX (XX.X) |
| Number of units/drinks per week | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| IQR | | XX.X |
| Min | | XX |
| Max | | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.7.2 Alcohol consumption (prior treatment groups)

The core population Page X of X

| | | Treatment-<br>experienced<br>(N=XX) | Naïve<br>(N=XX) |
|---|---|---|---|
| Alcohol use | | | |
| n | | XX | XX |
| Ex-drinker | n (%) | XX (XX.X) | XX (XX.X) |
| None | n (%) | XX (XX.X) | XX (XX.X) |
| Yes, occasional | n (%) | XX (XX.X) | XX (XX.X) |
| Yes, regular | n (%) | XX (XX.X) | XX (XX.X) |
| Number of units/drinks per week | | | |
| n | | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| IQR | | XX.X | XX.X |
| Min | | XX | XX |
| Max | | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.7.3 Alcohol consumption (treatment-experienced groups)

The core population Page X of X

| | | PEG-INF alpha (N=XX) | non-PEG-INF<br>alpha<br>(N=XX) | INF all (N=XX) | Ribavirin<br>(N=XX) |
|---|---|---|---|---|---|
| Alcohol use | | | | | |
| n | | XX | XX | XX | XX |
| Ex-drinker | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| None | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes, occasional | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes, regular | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Number of units/drinks per week | | | | | |
| n | | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X |
| IQR | | XX.X | XX.X | XX.X | XX.X |
| Min | | XX | XX | XX | XX |
| Max | | XX | XX | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).



AbbVie LLC P16-253 (CITRIN)

### Table 1.7.4 Alcohol consumption (Child Pugh score groups)

The core population Page X of X

| | | Score 5 (N=XX) | Score 6 (N=XX) |
|---------------------------------|-------|----------------|----------------|
| Alcohol use | | | |
| n | | XX | XX |
| Ex-drinker | n (%) | XX (XX.X) | XX (XX.X) |
| None | n (%) | XX (XX.X) | XX (XX.X) |
| Yes, occasional | n (%) | XX (XX.X) | XX (XX.X) |
| Yes, regular | n (%) | XX (XX.X) | XX (XX.X) |
| Number of units/drinks per week | | | |
| n | | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| IQR | | XX.X | XX.X |
| Min | | XX | XX |
| Max | | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.7.1, tables for the target and the safety populations will be constructed:

Table 1.7.5 Alcohol consumption Table 1.7.6 Alcohol consumption



## **Medical history**

AbbVie LLC P16-253 (CITRIN)

### Table 1.8.1 Liver and/or CHC related co-morbidities

The core population Page X of X

| System Organ Class<br>Preferred Term [1] | Total<br>(N=XX)<br>n (%) / E |
|---|---|
| Overall | XX (XX.X) / XX |
| System Organ Class 1<br>Preferred Term A<br>Preferred Term A | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |
| ••• | ••• |
| System Organ Class 2<br>Preferred Term C<br>Preferred Term D | XX (XX.X) / XX<br>XX (XX.X) / XX<br>XX (XX.X) / XX |
| ••• | |
| ••• | ••• |

N: the number of subjects in the core population. n: the number of subjects within a specific category. E: number of medical history events reported. Liver and/or chc related co-morbidities were coded using MedDRA 20.1. Percentages are calculated from the number of subjects in the core population. System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of Total frequency count.

[1] Within SOC patients may have reported more than one PT.



AbbVie LLC P16-253 (CITRIN)

### Table 1.8.2 Liver and/or CHC related co-morbidities (prior treatment groups)

The core population Page X of X

| System Organ Class<br>Preferred Term [1] | Treatment-experienced<br>(N=XX)<br>n (%) / E | Naïve<br>(N=XX)<br>n (%) / E |
|---|---|---|
| Overall | XX (XX.X) / XX | XX (XX.X) / XX |
| System Organ Class 1 | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX |
| ••• | ••• | • • • |
| System Organ Class 2 | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term C | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term D | XX (XX.X) / XX | XX (XX.X) / XX |
| • • • | ••• | ••• |
| | ••• | • • • |

N: the number of subjects in the core population. n: the number of subjects within a specific category. E: number of medical history events reported. Liver and/or chc related co-morbidities were coded using MedDRA 20.1. Percentages are calculated from the number of subjects in the core population. System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of Treatment-experienced frequency count.

[1] Within SOC patients may have reported more than one PT.



AbbVie LLC P16-253 (CITRIN)

### Table 1.8.2 Liver and/or CHC related co-morbidities (treatment-experienced groups)

The core population Page X of X

| System Organ Class<br>Preferred Term [1] | PEG-INF alpha<br>(N=XX)<br>n (%) / E | non-PEG-INF alpha<br>(N=XX)<br>n (%) / E | INF all (N=XX) n (%) / E | Ribavirin<br>(N=XX)<br>n (%) / E |
|---|---|---|---|---|
| Overall | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| System Organ Class 1 | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| • • • | • • • | • • • | • • • | • • • |
| System Organ Class 2 | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term C | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term D | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX | XX (XX.X) / XX |
| ••• | ••• | ••• | | • • • |
| | ••• | ••• | | • • • |

N: the number of subjects in the core population. n: the number of subjects within a specific category. E: number of medical history events reported. PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).

Liver and/or chc related co-morbidities were coded using MedDRA 20.1. Percentages are calculated from the number of subjects in the core population. System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of INF all frequency count.

[1] Within SOC patients may have reported more than one PT.



AbbVie LLC P16-253 (CITRIN)

### Table 1.8.2 Liver and/or CHC related co-morbidities (Child Pugh score groups)

The core population Page X of X

| System Organ Class<br>Preferred Term [1] | Score 5<br>(N=XX)<br>n (%) / E | Score 6<br>(N=XX)<br>n (%) / E |
|---|---|---|
| Overall | XX (XX.X) / XX | XX (XX.X) / XX |
| System Organ Class 1 | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term A | XX (XX.X) / XX | XX (XX.X) / XX |
| ••• | • • • | • • • |
| System Organ Class 2 | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term C | XX (XX.X) / XX | XX (XX.X) / XX |
| Preferred Term D | XX (XX.X) / XX | XX (XX.X) / XX |
| ••• | ••• | • • • |
| • • • | ••• | |

N: the number of subjects in the core population. n: the number of subjects within a specific category. E: number of medical history events reported. Liver and/or chc related co-morbidities were coded using MedDRA 20.1. Percentages are calculated from the number of subjects in the core population. System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of score 5 frequency count.

[1] Within SOC patients may have reported more than one PT.

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.8.1, tables for the target and the safety populations will be constructed:

Table 1.8.5 Liver and/or CHC related co-morbidities Table 1.8.6 Liver and/or CHC related co-morbidities



Similar to tables 1.8.X, tables for the other co-morbidities will be constructed:

for the core population

Table 1.9.1 Other co-morbidities

Table 1.9.2 Other co-morbidities (prior treatment groups)

Table 1.9.3 Other co-morbidities (treatment-experienced groups)

Table 1.9.4 Other co-morbidities (Child Pugh score groups)

for the target and safety populations

Table 1.9.5 Other co-morbidities Table 1.9.6 Other co-morbidities



### **Co-infections**

AbbVie LLC P16-253 (CITRIN)

### Table 1.10.1 Co-infections

The core population 

| Diagnosis | Total<br>(N=XX)<br>n (%) |
|-----------------------------------|--------------------------|
| Hepatitis B | XX (XX.X) |
| Human immunodeficiency virus(HIV) | XX (XX.X) |
| Tuberculosis | XX (XX.X) |
| Schistosomiasis | XX (XX.X) |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as (100 x n/N).

Program code, date, time Data extracted: DD.MM.YYYY

AbbVie LLC P16-253 (CITRIN)

### Table 1.10.2 Co-infections (prior treatment groups)

The core population 

| Diagnosis | Treatment-<br>experienced<br>(N=XX)<br>n (%) | Naïve<br>(N=XX)<br>n (%) |
|---|---|---|
| Hepatitis B | XX (XX.X) | |
| Human immunodeficiency virus(HIV) | XX (XX.X) | |
| Tuberculosis | XX (XX.X) | |
| Schistosomiasis | XX (XX.X) | |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as (100 x n/N).



AbbVie LLC

P16-253 (CITRIN)

### Table 1.10.3 Co-infections (treatment-experienced groups)

The core population 

| Diagnosis | PEG-INF alpha<br>(N=XX)<br>n (%) | non-PEG-INF alpha<br>(N=XX)<br>n (%) | INF all (N=XX) n (%) | Ribavirin<br>(N=XX)<br>n (%) |
|---|---|---|---|---|
| Hepatitis B | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Human immunodeficiency virus(HIV) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Tuberculosis | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Schistosomiasis | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).

Program code, date, time Data extracted: DD.MM.YYYY

AbbVie LLC P16-253 (CITRIN)

### Table 1.10.4 Co-infections (Child Pugh score groups)

The core population 

| Diagnosis | Score 5<br>(N=XX)<br>n (%) | Score 6<br>(N=XX)<br>n (%) |
|---|---|---|
| Hepatitis B | XX (XX.X) | XX (XX.X) |
| Human immunodeficiency virus(HIV) | XX (XX.X) | XX (XX.X) |
| Tuberculosis | XX (XX.X) | XX (XX.X) |
| Schistosomiasis | XX (XX.X) | XX (XX.X) |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as (100 x n/N).

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.10.1, tables for the target and the safety populations will be constructed:



Table 1.10.5 Co-infections
Table 1.10.6 Co-infections



AbbVie LLC P16-253 (CITRIN)

### Table 1.11.1 HIV most recent test results

The core population Page X of X

| | | Total<br>(N=XX) |
|------------------------------------|-------|-----------------|
| CD4 T-cell count | | (N-VV) |
| n | | XX |
| less 50 | n (%) | XX (XX.X) |
| 50-199 | n (%) | XX (XX.X) |
| 200-349 | n (%) | XX (XX.X) |
| 350-500 | n (%) | XX (XX.X) |
| >500 | n (%) | XX (XX.X) |
| HIV-RNA test | | |
| Result | | |
| n | | XX |
| undetectable | n (%) | XX (XX.X) |
| detectable | n (%) | XX (XX.X) |
| Below limit of quantification | | |
| n | | XX |
| Yes | n (%) | XX (XX.X) |
| No | n (%) | XX (XX.X) |
| Quantitative result (unit measure) | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.XX |
| Median | | XX.X |
| IQR | | XX.X |
| Min | | XX |
| Max | | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC P16-253 (CITRIN)

### Table 1.11.2 HIV most recent test results (prior treatment groups)

The core population Page X of X

| | | Treatment-<br>experienced<br>(N=XX)<br>n (%) | Naïve<br>(N=XX)<br>n (%) |
|---|---|---|---|
| CD4 T-cell count | | | |
| n | | XX | XX |
| less 50 | n (%) | XX (XX.X) | XX (XX.X) |
| 50-199 | n (%) | XX (XX.X) | XX (XX.X) |
| 200-349 | n (%) | XX (XX.X) | XX (XX.X) |
| 350-500 | n (%) | XX (XX.X) | XX (XX.X) |
| >500 | n (%) | XX (XX.X) | XX (XX.X) |
| HIV-RNA test | | | |
| Result | | | |
| n | | XX | XX |
| undetectable | n (%) | XX (XX.X) | XX (XX.X) |
| detectable | n (%) | XX (XX.X) | XX (XX.X) |
| Below limit of quantification | | | |
| n | | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) |
| Quantitative result (unit measure) | | | |
| n | | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| IQR | | XX.X | XX.X |
| Min | | XX | XX |
| Max | | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



AbbVie LLC

### P16-253 (CITRIN)

# Table 1.11.3 HIV most recent test results (Child Pugh score groups) The core population

Page X of X

| | | PEG-INF alpha<br>(N=XX) | non-PEG-INF alpha<br>(N=XX) | INF all (N=XX) | Ribavirin<br>(N=XX) |
|---|---|---|---|---|---|
| CD4 T-cell count | | | | | |
| n | | XX | XX | XX | XX |
| less 50 | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 50-199 | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 200-349 | n (응) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 350-500 | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| >500 | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| HIV-RNA test | | | | | |
| Result | | | | | |
| n | | XX | XX | XX | XX |
| undetectable | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| detectable | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Below limit of quantification | | | | | |
| n | | XX | XX | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Quantitative result (unit measure) | | | | | |
| n | | XX | XX | XX | XX |
| Mean | | XX.X | XX.X | XX.X | XX.X |
| SD | | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | | XX.X | XX.X | XX.X | XX.X |
| IQR | | XX.X | XX.X | XX.X | XX.X |
| Min | | XX | XX | XX | XX |
| Max | | XX | XX | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).



AbbVie LLC P16-253 (CITRIN)

### Table 1.11.4 HIV most recent test results (prior treatment groups)

The core population Page X of X

| | | Score 5 (N=XX) | Score 6 (N=XX) |
|------------------------------------|-------|----------------|----------------|
| CD4 T-cell count | | | |
| n | | XX | XX |
| less 50 | n (%) | XX (XX.X) | XX (XX.X) |
| 50-199 | n (%) | XX (XX.X) | XX (XX.X) |
| 200-349 | n (%) | XX (XX.X) | XX (XX.X) |
| 350-500 | n (%) | XX (XX.X) | XX (XX.X) |
| >500 | n (응) | XX (XX.X) | XX (XX.X) |
| HIV-RNA test | | | |
| Result | | | |
| n | | XX | XX |
| undetectable | n (%) | XX (XX.X) | XX (XX.X) |
| detectable | n (응) | XX (XX.X) | XX (XX.X) |
| Below limit of quantification | | | |
| n | | XX | XX |
| Yes | n (%) | XX (XX.X) | XX (XX.X) |
| No | n (%) | XX (XX.X) | XX (XX.X) |
| Quantitative result (unit measure) | | | |
| n | | XX | XX |
| Mean | | XX.X | XX.X |
| SD | | XX.XX | XX.XX |
| Median | | XX.X | XX.X |
| IQR | | XX.X | XX.X |
| Min | | XX | XX |
| Max | | XX | XX |

N: the number of subjects in the core population. n: the number of valid measurements. Percentages are calculated as  $(100 \times n/N)$ .



Similar to table 1.11.1, tables for the target and the safety populations will be constructed:

Table 1.11.5 HIV most recent test results Table 1.11.6 HIV most recent test results



### **Prior and concurrent medications**

AbbVie LLC P16-253 (CITRIN)

### Table 1.12.1 Prior Medications for CHC

The core population Page X of X

| Pharmacological subgroup WHODD chemical substance | Total<br>(N=XX)<br>n (%) /E |
|---|---|
| Total [1] | XX (XX.X) /XX |
| xxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX |
| ••• | ••• |
| xxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX |
| ••• | ••• |
| ••• | ••• |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . E: number of medical history events reported. Prior medications were coded using WHODD version Jun 2015. Each subject is only counted once per preferred name and once per ATC group. ATC group and preferred names within each ATC group are sorted in descending order of Total frequency count.

[1] The Total line displays the number (n) and the proportion (%) of patients, who have at least one prior medication prescription, and the total number of prior medication prescriptions.



AbbVie LLC

# P16-253 (CITRIN) Table 1.12.2 Prior Medications for CHC (prior treatment groups)

The core population Page X of X

| Pharmacological subgroup<br>WHODD chemical substance | Treatment-experienced (N=XX) n (%) / E | Naïve<br>(N=XX)<br>n (%) / E |
|---|---|---|
| Total [1] | XX (XX.X) /XX | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | |
| ••• | ••• | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | |
| ••• | • • • | |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . E: number of medical history events reported. Prior medications were coded using WHODD version Jun 2015. Each subject is only counted once per preferred name and once per ATC group. ATC group and preferred names within each ATC group are sorted in descending order of Treatment-experienced frequency count. [1] The Total line displays the number (n) and the proportion (%) of patients, who have at least one prior medication prescriptions, and the total number of prior medication prescriptions.



AbbVie LLC P16-253 (CITRIN)

### Table 1.12.3 Prior Medications for CHC (treatment-experienced groups)

The core population Page X of X

| Pharmacological subgroup WHODD chemical substance | PEG-INF alpha<br>(N=XX)<br>n (%) / E | non-PEG-INF alpha<br>(N=XX)<br>n (%) / E | INF all (N=XX) n (%) / E | Ribavirin<br>(N=XX)<br>n (%) / E |
|---|---|---|---|---|
| Total [1] | XX (XX.X) /XX | | | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX | | | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | | | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | | | |
| ••• | • • • | | | |
| xxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX | | | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX (XX.X) /XX | | | |
| ••• | ••• | | | |
| ••• | ••• | | | |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . PEG-INF alpha: Pegylated Interferon alpha. non-PEG-INF alpha: Interferon alpha (non-pegylated).

E: number of medical history events reported. Prior medications were coded using WHODD version Jun 2015. Each subject is only counted once per preferred name and once per ATC group. ATC group and preferred names within each ATC group are sorted in descending order of INF all frequency count.

<sup>[1]</sup> The Total line displays the number (n) and the proportion (%) of patients, who have at least one prior medication prescription, and the total number of prior medication prescriptions.



AbbVie LLC P16-253 (CITRIN)

#### Table 1.12.4 Prior Medications for CHC (Child Pugh score groups)

The core population Page X of X

| Pharmacological subgroup WHODD chemical substance | Score 5<br>(N=XX)<br>n (%) / E | Score 6<br>(N=XX)<br>n (%) / E |
|---|---|---|
| Total [1] | XX (XX.X) /XX | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX<br>XX (XX.X) /XX<br>XX (XX.X) /XX | |
| xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XX (XX.X) /XX<br>XX (XX.X) /XX | |
| | ••• | |

N: the number of subjects in the core population. n: the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . E: number of medical history events reported. Prior medications were coded using WHODD version Jun 2015. Each subject is only counted once per preferred name and once per ATC group. ATC group and preferred names within each ATC group are sorted in descending order of score 5 frequency count. [1] The Total line displays the number (n) and the proportion (%) of patients, who have at least one prior medication prescription, and the total number of prior medication prescriptions.

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 1.12.1, tables for the target and the safety populations will be constructed:

Table 1.12.5 Prior Medications for CHC Table 1.12.6 Prior Medications for CHC



Similar to tables 1.12.X, tables for the concurrent medications for CHC will be constructed:

for the core population

Table 1.13.1 Concurrent Medications for CHC
Table 1.13.2 Concurrent Medications for CHC (prior treatment groups)
Table 1.13.3 Concurrent Medications for CHC (treatment-experienced groups)
Table 1.13.4 Concurrent Medications for CHC (Child Pugh score groups)

for the target and safety populations

Table 1.13.5 Concurrent Medications for CHC Table 1.13.6 Concurrent Medications for CHC



### **Effectiveness Analyses (TP)**

AbbVie Ltd P16-253

### Table 2.1.1.1 Percentage for effectiveness endpoints

The target population (TP) Page X of X

| Parameter Statistics | Total<br>(N=XX)<br>n (%)<br>[95% CI] |
|---|---|
| SVR12 achieving (single last HCV RNA value <50 IU/mL 12 weeks after the last actual dose of the ABBVIE REGIMEN) | XX (XX.X)<br>[XX.XX - XX.XX] |
| SVR12 non-response | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with breakthrough (at least one documented HCV RNA value <50 IU/mL followed by HCV RNA ≧50 IU/mL during treatment) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Failure to suppress (each measured on-treatment HCV RNA value ≧50 IU/mL) | XX (XX.X) [XX.XX - XX.XX] |
| Patients with relapse (HCV RNA value <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA ≧50 IU/mL post-treatment) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with premature study drug discontinuation with no on-treatment virological failure (breakthrough or failure to suppress) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with missing SVR12 data | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with virological response (HCV RNA <50 IU/mL) at EoT | XX (XX.X)<br>[XX.XX - XX.XX] |

N: the number of subjects in the target population. n: number of subjects within a specific category. Percentages are calculated as  $100 \times (n/N)$ . EoT: end of treatment. SVR12: sustained virological response at 12 weeks after EoT. 95% CI: 95% confidence interval (the Clopper-Pearson method).



AbbVie Ltd P16-253

### Table 2.1.2.1 Percentage for effectiveness endpoints without patients with missing SVR12 results

The target population (TP)

Page X of X

| Parameter Statistics | Total<br>(N=XX)<br>n (%)<br>[95% CI] |
|---|---|
| SVR12 achieving (single last HCV RNA value <50 IU/mL 12 weeks after the last actual dose of the ABBVIE REGIMEN) | XX (XX.X)<br>[XX.XX - XX.XX] |
| SVR12 non-response | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with breakthrough (at least one documented HCV RNA value <50 IU/mL followed by HCV RNA ≧50 IU/mL during treatment) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Failure to suppress (each measured on-treatment HCV RNA value ≧50 IU/mL) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with relapse (HCV RNA value <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA $\geq$ 50 IU/mL post-treatment) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with premature study drug discontinuation with no on-treatment virological failure (breakthrough or failure to suppress) | XX (XX.X)<br>[XX.XX - XX.XX] |
| Patients with virological response (HCV RNA <50 IU/mL) at EoT | XX (XX.X)<br>[XX.XX - XX.XX] |

N: the number of subjects in the target population. n: number of subjects within a specific category. Percentages are calculated as  $100 \times (n/N)$ . EoT: end of treatment. SVR12: sustained virological response at 12 weeks after end of treatment. CI^ confidence interval. 95% confidence intervals calculated using the Clopper-Pearson method.



AbbVie LLC P15-743 (HCV RWE)

### Table 2.1.X.1 SVR12 achieving. Univariate logistic regression results

The core population Page X of X

| | Total |
|------------------------------|-----------------------|
| Predictor 1 | |
| Patients for analysis (n) | XXX |
| Convergence criterion status | xxxxxxxxxx |
| OR (95% Wald CI) | X.XXX (X.XXX - X.XXX) |
| p-value | 0.xxxx |
| Predictor 2 | |
| Patients for analysis (n) | XXX |
| Convergence criterion status | xxxxxxxxxx |
| Reference level | xxxxxxxxxx |
| OR (95% Wald CI) for Level X | X.XXX (X.XXX - X.XXX) |
| p-value for Male | 0.xxxx |

SVR12: sustained virological response at 12 weeks after end of treatment. OR: odds ratio. CI: confidence interval.



AbbVie LLC P15-743 (HCV RWE)

#### Table 2.1.X.2 SVR12 achieving. Multiple logistic regression results

The core population Page X of X

| | Overall |
|---------------------------|-----------------------|
| Patients for analysis (n) | XXX |
| Predictor 1 | |
| OR (95% Wald CI) | X.XXX (X.XXX - X.XXX) |
| p-value | 0.XXXX |

SVR12: sustained virological response at 12 weeks after end of treatment. OR: odds ratio. CI: confidence interval.

Program code, date, time

Data extracted: DD.MM.YYYY

Similar to table for SVR12 achieving univariate logistic regression results, tables for the following variables (outcomes) will be constructed (if applicable):

Table 2.1.X.1 Virological response at EoT. Univariate logistic regressions results Table 2.1.X.2 Virological response at EoT. Multiple logistic regression results

Table 2.1.X.1 Relapse after EoT. Univariate logistic regressions results
Table 2.1.X.2 Relapse after EoT. Multiple logistic regression results



### **Effectiveness Analyses (CP)**

Similar to tables 2.1.1.X-2.1.2.X, the following tables will be constructed for the core population:

Table 2.2.1.1 Percentage for effectiveness endpoints
Table 2.2.2.1 Percentage for effectiveness endpoints without patients with missing SVR12 results

Similar to tables 2.1.X.1-2.1.X.2, tables for the following variables (outcomes) will be constructed (if applicable) for the core population:

Table 2.2.X.1 SVR12 achieving. Univariate logistic regression results Table 2.2.X.2 SVR12 achieving. Multiple logistic regression results

Table 2.2.X.1 Virological response at EoT. Univariate logistic regressions results Table 2.2.X.2 Virological response at EoT. Multiple logistic regression results

Table 2.2.X.1 Relapse after EoT. Univariate logistic regressions results
Table 2.2.X.2 Relapse after EoT. Multiple logistic regression results



### **Effectiveness Analyses (CPSFU)**

Similar to tables 2.1.1.X-2.1.2.X, the following tables will be constructed for the core population with sufficient follow-up data (CPSFU):

Table 2.3.1.1 Percentage for effectiveness endpoints (main analysis)
Table 2.3.2.1 Percentage for effectiveness endpoints without patients with missing SVR12 results (main analysis)

Similar to tables 2.1.X.1-2.1.X.2, tables for the following variables (outcomes) will be constructed (if applicable) for the core population:

Table 2.3.X.1 SVR12 achieving. Univariate logistic regression results Table 2.3.X.2 SVR12 achieving. Multiple logistic regression results

Table 2.3.X.1 Virological response at EoT. Univariate logistic regressions results Table 2.3.X.2 Virological response at EoT. Multiple logistic regression results

Table 2.3.X.1 Relapse after EoT. Univariate logistic regressions results
Table 2.3.X.2 Relapse after EoT. Multiple logistic regression results



**Exposure** 

AbbVie LLC P16-253 (CITRIN)

### Table 3.1 AbbVie REGIMEN intake

The safety population Page X of X

| | Total (N = XX) |
|-----------------------------------------------------------|----------------|
| Actual duration ABBVIE REGIMEN [1] | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| Subjects with collected deviating duration reasons | XX (XX.X) |
| Reasons for deviating duration: | |
| AE or SAE (Physician decision) | XX (XX.X) |
| Virological non-response (Physician decision) | XX (XX.X) |
| Rebound or breakthrough (Physician decision) | XX (XX.X) |
| Resistance to DAA (Physician decision) | XX (XX.X) |
| Patient refused to continue treatment | XX (XX.X) |
| Patient withdrew consent to participate in the study | XX (XX.X) |
| Lost to follow-up | XX (XX.X) |
| ••• | ••• |
| PARITAPREVIR/R-OMBITASVIR | |
| Subjects with intake missing for at least 7 days in a row | XX (XX.X) |
| Percentage of target dose taken (%) Weeks 1-4 | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| Weeks 5-8 | |
| n | XX |
| Mean | XX.X |
| Data MATRIX Ltd. | Page 65 of 79 |



| SD | XX.XX |
|-----------------------------------------------------------|-----------|
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| Weeks 9-12 | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| DASABUVIR | |
| Subjects with intake missing for at least 7 days in a row | XX (XX.X) |
| Percentage of target dose taken (%) | |
| Weeks 1-4 | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| Weeks 5-8 | |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| Min | XX |
| Max | XX |
| Weeks 9-12 | m |
| n | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| IQR | XX.X |
| ngk<br>Min | XX XX |
| Min<br>Max | XX<br>XX |
| I <sup>VI</sup> d X | X X |

N: the number of subjects in the target population.

n: the number of subjects within a specific category. Percentages were calculated as (100 x n/N).

<sup>[1]</sup> This parameter is calculated as interval (in days) between date of first intake and date of last intake of treatment.



### Adverse events

AbbVie LLC P16-253 (CITRIN)

#### Table 3.2.1 Adverse events

The safety population Page X of X

| System organ class (SOC) Preferred term (PT) | Total<br>(N=XX)<br>n (%) /E |
|---|---|
| Total [1] | XX (XX.X) /XX |
| System organ class 1 Preferred term A | XX (XX.X) /XX<br>XX (XX.X) /XX |
| Preferred term B | ••• |
| | ••• |
| System organ class 2 | |
| ••• | ••• |
| | ••• |

N: the number of patients in the safety population.

Similar to table 3.2.1, table 3.2.2 will be constructed:

Program code, date, time

Data extracted: DD.MM.YYYY

n: the number of patients who have AE with appropriate SOC/PT. Percentages are calculated as  $(100 \times n/N)$ .

E: the number of AE episodes, which have an appropriate SOC and/or PT.

Patients with several AEs having the same SOC and PT are accounted only once for appropriate SOC and PT.

<sup>[1]</sup> The Total line displays the number (n) and the proportion (%) of patients who have at least on AE as well as the total number of AE episodes in the study.

The coding is carried out by the dictionary MedDRA v.20.0.

The table does not include AEs that occurred prior to the first intake of the study drug.

The data is sorted alphabetically: first by SOC, then by PT.



Table 3.2.2 Serious adverse events



AbbVie LLC P16-253 (CITRIN)

### Table 3.2.3 Adverse events by relationship to the study drug

The safety population

Page X of X

| System Organ Class (SOC) Preferred term (PT) | Relationship<br>to the study drug | Total<br>(N=XX)<br>n (%) /E |
|---|---|---|
| Total [1] | Reasonable possibility<br>No reasonable possibility | XX (XX. X) /XX<br>XX (XX. X) /XX |
| | Total | XX (XX.X) /XX |
| System Organ Class 1 | Reasonable possibility<br>No reasonable possibility<br>Total | XX (XX.X) /XX<br>XX (XX.X) /XX<br>XX (XX.X) /XX |
| Preferred term A | Reasonable possibility<br>No reasonable possibility<br>Total | XX (XX.X) /XX<br>XX (XX.X) /XX<br>XX (XX.X) /XX |
| Preferred term B | Reasonable possibility | XX (XX.X) /XX |
| System Organ Class 2 | Reasonable possibility | XX (XX.X) /XX |

N: the number of patients in the safety population.

Each SOC/PT category includes only AEs with the highest relationship to the study drug in each patient. Each patient is counted only once in the Total lines and in the lines for each SOC or SOC/PT categories. Thus, if patient has several AEs with the same SOC and PT but different relationship to the drug, only the AEs with maximum relashionship will be accounted, while each patient will be accounted only once in line which corresponds the highest relationship of his AEs.

[1] The Total lines displays the number (n) and the proportion (%) of patients who have AEs. Each patient is counted once in line which corresponds the highest relationship of all his AEs. #E displays the number of all AEs episodes with appropriate relationship to the drug in the study.

The coding is carried out by the dictionary MedDRA v.20.0. The table does not include AEs that occurred prior to the first intake of the study drug.

The data is sorted alphabetically: first by SOC, then by PT and relationship to the drug.

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 3.2.3, table 3.2.4 will be constructed:

n: the number of patients who have AE with appropriate SOC/PT. Percentages are calculated as (100 x n/N).

E: the number of AE episodes, which have an appropriate SOC and/or PT.



Table 3.2.4 Serious adverse events by relationship to the study drug



AbbVie LLC P16-253 (CITRIN)

### Table 3.2.5 Adverse events by severity

The safety population Page X of X

| System Organ Class (SOC) Preferred term (PT) | Severity | Total<br>(N=XX)<br>n (%) /E |
|---|---|---|
| Total [1] | Severe | XX (XX.X) /XX |
| | Moderate | XX(XX.X) /XX |
| | Mild | |
| | Total | XX(XX.X) /XX |
| System Organ Class 1 | Severe | XX(XX.X) /XX |
| | Moderate | XX (XX.X) /XX |
| | Mild | |
| | Total | XX (XX.X) /XX |
| Preferred term A | Severe | XX (XX.X) /XX |
| | Moderate | XX (XX.X) /XX |
| | Mild | |
| | Total | XX(XX.X) /XX |
| Preferred term B | Consens | VV (VV V) /VV |
| | Severe | XX(XX.X) /XX |
| | Moderate | XX(XX.X) /XX |
| | Mild | |
| | Total | XX (XX.X) /XX |
| | | ••• |
| System Organ Class 2 | Severe | XX(XX.X) /XX |
| | Moderate | XX (XX.X) /XX |



| System Organ Class (SOC) Preferred term (PT) | Severity | Total<br>(N=XX)<br>n (%) /E |
|---|---|---|
| | Mild | |
| | Total | XX(XX.X) /XX |
| ••• | •••• | |
| ••• | ••• | ••• |

N: the number of patients in the safety population.

Each SOC/PT category includes only AEs with the highest severity in each patient. Each patient is counted only once in the Total lines and in the lines for each SOC or SOC/PT categories. Thus, if patient has several AEs with the same SOC and PT but different severity, only the AEs with maximum severity will be accounted, while each patient will be accounted only once in line which corresponds the highest severity of his AEs.

[1] The Total lines displays the number (n) and the proportion (%) of patients who have AEs. Each patient is counted once in line which corresponds the highest severity of all his AEs. #E displays the number of all AEs episodes with appropriate severity in the study.

The coding is carried out by the dictionary MedDRA v.20.0.

The table does not include AEs that occurred prior to the first intake of the study drug.

The data is sorted alphabetically: first by SOC, then by PT and relationship to the drug.

Program code, date, time Data extracted: DD.MM.YYYY

Similar to table 3.2.5, table 3.2.6 will be constructed:

Table 3.2.6 Serious adverse events by severity

n: the number of patients who have AE with appropriate SOC/PT. Percentages are calculated as  $(100 \times n/N)$ .

E: the number of AE episodes, which have an appropriate SOC and/or PT.



# Hematology

AbbVie LLC P16-253 (CITRIN)

### Table 3.3.1 Hematology. Descriptive statistics

The safety population Page X of X

| Parameter<br>Visit<br>Statistics | Total (N = XX) | Change from baseline $(N = XX)$ |
|---|---|---|
| Hemoglobin (unit measure) | | |
| Visit 1 | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.XX | |
| Median | XX.X | |
| IQR | XX.X | |
| Min | XX | |
| Max | XX | |
| EoT | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| IQR | XX.X | XX.X |
| Min | XX | XX |
| Max | XX | XX |
| SVR12 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| IQR | XX.X | XX.X |
| Min | XX | XX |



| Parameter<br>Visit<br>Statistics | Total (N = XX) | Change from baseline $(N = XX)$ |
|---|---|---|
| Max | XX | XX |
| Platelets (unit measure) | | |
| Prothrombin time (unit measure) | | |
| ••• | | |

N: the number of patients in the safety population.

IQR: interquartile range.

EoT: end of treatment.

SVR12: sustained virological response at 12 weeks after end of treatment.

Table displays descriptive statistics for general blood test parameters values and their changes from baseline (visit 1).

n: the number of valid measurements.

SD: standard deviation.



AbbVie LLC P16-253 (CITRIN)

### Table 3.3.2 Hematology. Clinical assessments

The safety population Page X of X

| Parameter | m 1 |
|--------------|-----------|
| Visit | |
| Value | · · · |
| Hemoglobin | |
| Visit 1 | |
| n | XXX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| EoT | |
| n | XXX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| SVR12 | |
| n | XXX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |



| Visit<br>Value | Total $(N = XX)$ |
|----------------|------------------|
| Platelets | |
| ••• | |

N: the number of patients in the safety population.

n: the number of valid measurements. Percentages are based on the number of valid measurements at analyzed visit.

CS: clinically significant.

NCS: not clinically significant.

EoT: end of treatment.

Prothrombin time

Parameter

SVR12: sustained virological response at 12 weeks after end of treatment.



AbbVie LLC P16-743 (CITRIN)

### Table 3.3.3 Hematology. Shift table

The safety population Page X of X

| arameter | | Baseline ( | visit 1) | |
|----------------|-----------|--------------|-------------|----------------|
| Visit<br>Value | Normal | Abnormal NCS | Abnormal CS | Total assessed |
| emoglobin | | | | |
| Visit 1 | | | | |
| Normal | | | | XX (XX.X) |
| Abnormal NCS | | | | XX (XX.X) |
| Abnormal CS | | | | XX (XX.X) |
| Total assessed | | | | XX (100) |
| ЕоТ | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal NCS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal CS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total assessed | XX (100) | XX (100) | XX (100) | XX (100) |
| SVR12 | | | | |
| Normal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal NCS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Abnormal CS | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total assessed | XX (100) | XX (100) | XX (100) | XX (100) |

Platelets

 Data MATRIX Ltd.



| Parameter | Baseline (visit 1) | | | |
|---|---|---|---|---|
| Visit | Normal | Normal NCS | Abnormal CS | Total assessed |
| Value | | | | |
| Prothrombin time | | | | |

CS: clinically significant.

NCS: not clinically significant.

EoT: end of treatment.

SVR12: sustained virological response at 12 weeks after end of treatment.

Percentages are based on the number of patients with a non-missing assessment on time point and on baseline (visit 1).



## **Blood chemistry**

Similar to tables 3.3.1-3.3.3, the following tables will be constructed:

Table 3.4.1 Blood chemistry. Descriptive statistics
Table 3.4.2 Blood chemistry. Clinical assessments
Table 3.4.3 Blood chemistry. Shift table